CLINICAL TRIAL: NCT02316483
Title: Genetic Contribution to the Pathophysiology of the Charcot Foot in Qatari Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Other Study IDs: 13-00031 [JIRB]
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Charcot Arthropathy; Type 2 Diabetes
MeSH Terms: conditions — Arthropathy, Neurogenic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group I: T2D and Charcot foot: Individuals with confirmed diagnosis of type 2 diabetes, using the American Diabetes Association guidelines and confirmed diagnosis of Charcot foot, based on clinical and radiological evidence of Charcot foot.
- Group II: T2D neuropathy, no charcot: Individuals with type 2 diabetes and presence of neuropathy but the absence of Charcot foot.
- Group III: Control, non-diabetic: Individuals without history of type 2 diabetes.

SUMMARY:
To assess the hypothesis that Charcot foot is associated with more vascular complications compared to matched diabetic patients without Charcot foot and to classify patients with Charcot foot according to the human genetic classification of the Qatari population.

DETAILED DESCRIPTION:
Diabetes is a serious health issue for the Qatari population since approximately 1/5 of the population has Type 2 Diabetes, which is 2-3 times higher than the world average. Although much of the clinical studies of diabetes often focused on microvascular phenotypes such as retinopathy and nephropathy, and macrovascular diseases presenting clinically as myocardial infarction, stroke, and peripheral vascular disease, other rare complications such as Charcot foot disease confer a significant burden in Qatar diabetic population, leading to decreased life quality.

Charcot foot is estimated to affect 0.8% to 8% of diabetic populations. It occurs most commonly in patients with diabetes complicated by severe peripheral neuropathy, often with coexisting sympathetic denervation, causing increased blood flow to the foot and increased bone resorption.

Uncontrolled and inappropriate inflammation leading to bone resorption and deformation has been the hallmark of diabetic Charcot foot pathophysiology. There are two major theories that provide the likely mechanism of the disease. The "neurovascular (French) theory" suggests that increased blood flow, as a result of autonomic neuropathy, can lead to bone destruction and mechanical debilitation. On the other hand, the "neurotraumatic (German) theory" argues that the loss of protective sensation leads to unperceived injury and trauma in the insensate foot. One can argue that the pathogenesis of Charcot neuro-arthropathy is most likely a combination of these processes. For unknown reasons, Charcot foot is trigged only in some susceptible individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide informed consent
2. Must hold Qatari passport
3. Males or Females ages 30 years or older to minimize the potential confounding contribution of other forms of diabetes mellitus
4. In patients with Diabetes, no concomitant diseases except for micro- and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome (hypertension, dyslipidemia and obesity).
5. Not taking any chronic medications (except of the diabetes, cardiovascular related drugs, anti-inflammatory drugs and/or any other treatment used for Charcot foot).

Exclusion Criteria:

1. Other forms of diabetes (Type I, MODY, secondary diabetes)
2. Active pregnancy
3. Active infection or acute illness of any kind (except for Charcot foot)
4. Chronic inflammation (auto-immune diseases) or infection
5. Evidence of malignancy within the past 5 years
6. Chronic hematological disorders known to affect HBA1C results such as hemoglobinopathies (e.g., sickle cell disease and thalassemia), increased red-cell turnover (e.g., hemolytic anemia and spherocytosis)
7. Acute or critical limb ischemia.
8. Osteomyelitis
9. History of recent (within 6 months) immunosuppressive treatment including corticosteroids and anti-TNF-alpha compounds.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited for the study at Hamad Medical Corporation. Most of the subjects will belong to the oupatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-12; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Charcot Foot's vascular complications | 6 months
  Assess the hypothesis that Charcot Foot is associated with more vascular complications compared to match diabetic patients without Charcot foot
Charcot foot in monocyte epigenetics | 6 months
  Assess the hypothesis that Charcot foot disease reflects differences in monocyte epigenetics compared to other controls, particularly in genes involved in inflammation.
Assess the effect of initial methylation on kidney function in patients with type 2 diabetes mellitus, weather they have or not Charcot foot disease and for whom we have baseline kidney function, in a 2-year follow-up. | 6 months
HBA1C >8.5% on total and gene-specific methylation. | 6 months
  Assess the effect of improving diabetes control in patients with type 2 diabetes (Charcot foot and non-charcot foot patients) and a HBA1C >8.5% on total and gene-specific methylation.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Abi Khalil, MD, Principal Investigator — Weill Cornell Medical College in Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
All results of the proposed studies will be published in international peer-reviewed scientific journals, presented at meetings in Qatar, the regional and international conferences, and disseminated through the local Qatari media, seminars and lectures for high school and college students. The original data will be available to interested investigators using the conventional standards of biomedical science.

REFERENCES:
- [Derived] Pasquier J, Ramachandran V, Abu-Qaoud MR, Thomas B, Benurwar MJ, Chidiac O, Hoarau-Vechot J, Robay A, Fakhro K, Menzies RA, Jayyousi A, Zirie M, Al Suwaidi J, Malik RA, Talal TK, Najafi-Shoushtari SH, Rafii A, Abi Khalil C. Differentially expressed circulating microRNAs in the development of acute diabetic Charcot foot. Epigenomics. 2018 Oct;10(10):1267-1278. doi: 10.2217/epi-2018-0052. Epub 2018 Jun 5. PMID 29869523